CLINICAL TRIAL: NCT02083497
Title: COMPARISON BETWEEN RIGID FUNCTIONAL AND ELASTIC BANDAGE FOR STABILIZING ANKLE SUPPORT DURING THE MEMBER OF THE CHUTE FOOTBALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20559113.0.0000.5503
Record Dates: First submitted 2014-02-28; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Female Soccer Athletes
Keywords: kick; taping; dynamic equilibrium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No banding (Experimental): The volunteers who make up this group, held 18 kicks, 9 with the dominant leg and 9 with the non-dominant lower limb, without the intervention of any kind of bandage.
  Interventions: Other: without the use of banding
- Group with Rigid Bandage (Experimental): Volunteers carry out the same protocol described above, however, using rigid bandage. The bandage will be used for tape, Cremer brand and will be applied ankle support member of the individual, in order to limit the movement of the joint inversion.
  Interventions: Other: rigid bandage
- Group with elastic bands (Experimental): The protocol will be maintained, however, a brand elastic bandage Kinesio Sport applied to the lower support member of the individual, also in order to limit the movement of the joint inversion is used.
  Interventions: Other: elastic bands

INTERVENTIONS:
Other: rigid bandage
  Arms: Group with Rigid Bandage
Other: elastic bands
  Arms: Group with elastic bands
Other: without the use of banding
  Arms: No banding

SUMMARY:
To evaluate the influence of different types of ankle taping in dynamic equilibrium and the electrical activity of the support member during the sporting gesture kicking muscles.

DETAILED DESCRIPTION:
The most popular sport worldwide is football and there is, therefore , interest in detecting factors that may interfere with their practice. These factors are already investigated in the literature , in particular kick, gesture performed frequently , whereas in most situations is through him that achieves the main goal: to score. For this particular effort is needed balance to run it , and based on this body balance the ankle joint , responsible for the sense of position and movement of the body . Any deficit in the joint may interfere with the functional performance of the individual. The football players can use rigid or elastic bandages to prevent and optimize its performance . The use of bandages in different conditions is being studied , however analyzes performed during sporting gestures are scarce . Therefore , this study aims to evaluate the influence of two types of bandage ankle dynamic balance and activity power of the support limb during kicking through biomedical instrumentation muscles . Participate in the study 180 individuals practicing football , where half will consist of professional athletes and half will consist of sedentary individuals who have committed the sport of football at some point in life, aged 20 and 35 years of both sexes . All will perform the task of controlled shot on a force platform with one foot . Electrical activity through electromyography superfíciedos long and short fibular muscles , tibialis anterior and gluteus medius is collected.

The Gesture Controlled Shooting ( GCC ) will consist of the following phases :

* At the signal of the researcher , the individual should go to the center of the platform and reach , stand on one foot for execution of the kick, whereupon the cycle throughout the GCC ;
* After shooting the ball vertically , the participant will expect it to reach the maximum height and during the descent of the ball, run the kick with the member that is not supported on the platform , and the same shall be held at a convenient time for hit the target ;
* The effort must be made to the medial region of the foot ;
* The goal of the task is to hit the ball on target , accurately ;
* After foot contact with the ball for the execution of the kick, the individual should remain with leg support with visual focus directed to the target until the moment the search signal for it to leave the platform with the foot that held the kick and following with the foot that was in contact with the force platform ;
* Cycle the task will be completed .

  18 kicks will be performed, and 9 will be with the dominant leg and 9 with the non-dominant lower limb in each of the following situations : without bandage , bandage with rigid and elastic bandage .

To analyze the data , will be used ANOVA test for a significance level of 5 % . After the tests , the correlation is also carried out Pearson between the data obtained in the three situations of shooting . Therefore it is expected that the dynamic balance and muscle activation is influenced positively with the use of different types of taping , possibly showing what kind of application is most effective for use the sport of football.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who do not have a history of ligament surgery, intra-articular or muscular in the lower limbs;
* Individuals who do not have a history of ankle sprain;
* Individuals who have not suffered any muscle, ligament or intra-articular injury in the last six months;
* Be athlete of the sport of football.

Exclusion Criteria:

* Individuals who report having allergies to the material used in bandages;
* Individuals who have global ligamentous laxity.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
muscle electrical activity of the support member | individuals will be monitored during the task execution (9 kicks with each member), which gives an average of 3 hours.
  Muscle electrical activity of a member of support will be measured only during the time of the kicks, by surface electromyography (EMG), assessing rather the effect of intervention chosen at the time of the shooting sports gesture.

SECONDARY OUTCOMES:
dynamic equilibrium of the support limb in standing position | individuals will be monitored during the task execution (9 kicks with each member), which gives an average of 3 hours.
  The dynamic equilibrium of lower limb support will be measured only during the runtime of the chutes, through the force platform, assessing rather the effect of intervention chosen in the balance of the participant at the time of the shooting sports gesture.

OTHER OUTCOMES:
Number of hits on target shooting | an average of 3 hours
  The number of hits the target will be recorded during the activity execution (9 kicks).

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Engineering Laboratory of Sensory Motor, São José dos Campos, São Paulo, Brazil